CLINICAL TRIAL: NCT02273310
Title: Families Taking Control (FTC): Family-based Problem-solving Intervention for School-age Children With Sickle Cell Disease
Brief Title: Families Taking Control (FTC): Family-based Problem-solving Intervention for Children With Sickle Cell Disease
Acronym: FTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Drexel University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U54HL070585 (NIH); U54HL070585 (NIH)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Families Taking Control (Experimental): Families participate in a 1 day Problem-Solving Skills training for disease management intervention
  Interventions: Behavioral: Problem-Solving Skills Training for Disease Management
- Delayed Intervention Control (No Intervention): Families are given the opportunity to complete the Problem-solving Skills training for disease management intervention after assessment time 2.

INTERVENTIONS:
Behavioral: Problem-Solving Skills Training for Disease Management — Children and caregivers participated in a multi-family group to learn problem-solving skills as applied to disease management and school functioning in the context of sickle cell disease.
  Arms: Families Taking Control

SUMMARY:
This study aims to develop an effective, brief, family-based intervention targeting quality of life and school functioning for youth with sickle cell disease. Utilizing a randomized, delayed control group intervention methodology, the present study will systematically document the effectiveness of a family-based, one-day intervention plus booster phone calls to improve quality of life and increase school functioning for children with sickle cell disease transitioning to school and their families.

DETAILED DESCRIPTION:
Families Taking Control-School-age Intervention (FTC) will provide education and problem solving training for disease management and school functioning. In 4 sessions offered over the course of one day, families (patient, caregivers, and school-age siblings) will work together and individually to learn and apply the problem solving skills training model to relevant examples and family-specific problems, culminating in an outline of family goals to target after the intervention. The three booster phone calls will provide support to families in implementing the problem-solving model by addressing and refining goals and trouble-shooting barriers to implementation. Children and caregivers completed measures at baseline (prior to intervention participation) and 6 months later.

ELIGIBILITY:
Inclusion Criteria: English speaking, treated at one of two participating Sickle Cell Centers -

Exclusion Criteria: severe developmental delay or children/caregivers with severe psychopathology that would adversely affect their ability to participate

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Barakat, Ph.D., Principal Investigator — The Children's Hospital of Philadelphia/University of Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Families Taking Control: Families participate in a 1 day problem solving skills training intervention
  Problem Solving Training for Disease Management
- Delayed Intervention Control: Families are given the opportunity to complete the problem solving skills training intervention after assessment time 2.
Period: Overall Study
Arm/Group | Families Taking Control | Delayed Intervention Control
Started | 42 | 41
Completed | 24 | 38
Not Completed | 18 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Families Taking Control | Delayed Intervention Control | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.29 (2.12) | 8.66 (2.10) | 8.47 (2.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Child-Reported Health Related Quality of Life-School Functioning Subscale
Description: Assessed using the Pediatric Quality of Life Inventory, Scores range from 0-100 with higher scores indicating better quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Families Taking Control | Delayed Intervention Control
Number analyzed (Participants) | 24 | 38
units on a scale | 60.40 (23.89) | 64.60 (16.94)

2. Secondary Outcome: School Functioning-Absences
Description: School Absences reported by caregivers, Caregivers reported absences categorically (0-7 days = 1, 7-14 days = 2, etc). Higher numbers indicate more absences.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Weeks (1 week = 7 days)
Arm/Group | Families Taking Control | Delayed Intervention Control
Number analyzed (Participants) | 24 | 38
Weeks (1 week = 7 days) | 0.48 (0.77) | 1.10 (1.03)

3. Secondary Outcome: Number of Accommodations Provided to Families by Schools
Description: Number of Accommodations Provided to Families by Schools As reported by caregivers
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of Accommodations
Arm/Group | Families Taking Control | Delayed Intervention Control
Number analyzed (Participants) | 24 | 38
Number of Accommodations | 1.44 (1.35) | 1.38 (1.17)

4. Secondary Outcome: Acceptability of Intervention
Description: Families in the FTC group rated acceptability of participating in the intervention workshop. This measure was completed at the workshop (between baseline and 6 month assessments). This measure utilized a 5-point Likert-type scale (with the possible range of scores as 1-5), with higher scores indicating more positive feedback. Individual item scores are presented here. Participant results indicated a range of scores from from 2-5.
Time Frame: post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Families Taking Control
Number analyzed (Participants) | 28
units on a scale
  Caregiver-Interesting | 4.71 (0.46)
  Caregiver-Useful | 4.36 (0.68)
  Child-Interesting | 4.71 (0.85)
  Child-Useful | 4.39 (1.17)

ADVERSE EVENTS:
Arm/Group | Families Taking Control | Delayed Intervention Control
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No